CLINICAL TRIAL: NCT05804019
Title: Interventions Focusing on Nutrition and Physical Activities for Overweight and Obese Older Adults in Nursing Homes "IFEBO"
Brief Title: Nutritional and Physical Activities for Overweight and Obese Older Adults
Acronym: IFEBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Absalon (Other)
Collaborators: Odsherred, Denmark (Unknown); University of Copenhagen (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IFEBO; 1155-00001B (Other Grant/Funding Number: Innovation Fund Denmark); 2022-03 Tenna Christoffersen (Other Grant/Funding Number: Steno Diabetes Center Zealand)
Record Dates: First submitted 2023-03-01; First posted 2023-04-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Overweight, Obesity and Other Hyperalimentation
Keywords: Geriatric; Overnutrition; Physical function; Quality of Life
MeSH Terms: conditions — Overweight; Obesity; Overnutrition

STUDY DESIGN:
Intervention Model Description: Two arms (Nutritional and Physical Activity Intervention Group and Usual Care Group). Approximately 100 participants will be included and cluster randomized by the nursing home to either 6 months of nutritional and physical interventions or 6 months of usual care (control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Control) (No Intervention): Approximately 100 participants will be included and cluster randomized by nursing home (n= 3) to either 12 months of nutritional and physical intervention or 12 months of usual care (control). Usual Care Group will receive the usual care at the control nursing homes (n=3)
- Nutritional and Physical Intervention Group (Intervention Group) (Experimental): Approximately 100 participants will be included and cluster randomized by nursing home (n= 3) to either 12 months of nutritional and physical intervention or 12 months of usual care (control). The Nutritional and Physical Intervention Group will receive nutritional and physical interventions collaboratively defined by residents, relatives, care staff, and nursing home management during the PDSA workshops.
  Interventions: Behavioral: Nutritional and physical interventions

INTERVENTIONS:
Behavioral: Nutritional and physical interventions — The intervention is developed with a focus on nutritional needs and physical activities. The Plan-Do-Study-Act (PDSA) model is used to redefine issues and relevant actions together with residents, relatives, care staff, and nursing home management. The intervention will be developed based on new knowledge from sub-study 1, previous studies, practical experiences, the participant's experiences and wishes as well as the staff's experiences and wishes. Together they will form an implementation catalog, from here, the intervention nursing homes can select a relevant number of components, which will be tested and implemented in practice. The implementation duration is 6 months and the PDSA model is repeated at two-month intervals to strengthen and qualify the intervention. The PDSA model is known to the city's staff in advance and is additionally used in connection to continuing education. The Usual Care Group will continue the usual care.
  Arms: Nutritional and Physical Intervention Group (Intervention Group)

SUMMARY:
This cluster randomized trial aims to test nutritional and physical activity interventions in older adults in nursing homes. The overall research question are:

o What are the effects of nutritional and physical activity interventions on muscle function and quality of life in older adults with overweight and obesity? Participants' data on body composition, physical function, and diseases will be collected. Furthermore, participants will be interviewed for a questionnaire on quality of life and nutritional intake.

Researchers will compare three intervention nursing homes with three control nursing homes to see if nutrition and physical interventions have on physical function and quality of life.

DETAILED DESCRIPTION:
Background: The aging population is increasing both globally and nationally in Denmark. Concurrent with the generally rapidly increasing incidence of being overweight, a large number of older people risk facing several health problems associated with being overweight and obesity (Ow/O). Aging related to malnutrition or undernutrition has received a lot of attention. However, overnutrition described as Ow/O is also classified as a nutritional disorder or a nutrition-related condition, in the same term as malnutrition.

Today, all older adults in Danish nursing homes are offered an enriched diet type for malnourished older adults, focused on energy-dense snacks and a high-fat percentage. This is not necessarily an appropriate diet, but it is unknown which nutritional interventions are effective in maintaining/ improving physical functioning, independence, and quality of life. One of the concerns is that many older adults with Ow/O may have a loss of muscle mass, which can worsen with weight loss if this is not taken into account in the nutritional intervention. There is therefore a clear need to develop targeted interventions for older adults with Ow/O that can maintain or improve physical functioning and quality of life.

However, a literature review of interventions within the last 10 years shows that none of the interventions are aimed at healthy older adults ≥ 65 years with a BMI≥ 25kg/m2 and good physical functioning. Instead, interventions targeted older adults with Ow/O with either low physical functioning or chronic diseases. These interventions show that older adults can lose weight, but without significant positive effects on functioning and quality of life. The interventions in the studies contain complex nutrition and exercise interventions, and the differences in the intervention descriptions and target groups make it difficult to compare and point to safe and effective interventions. In addition, the studies show that there is no difference between whether the nutrition intervention applies to weight loss or weight maintenance interventions.

However, the above literature review has confirmed that there are older people with Ow/O, especially those with both low physical function and chronic disease, who may benefit from a nutritional intervention, which has led to a proposed approach. The characterization according to the screening model will be performed in sub-study 1 (a cross-sectional study) and adapted to be easy to use in a community health care setting.

In this trial, based on a descriptive pre-study, the project, in collaboration with the older adults, the care staff, and the project participants, developed and tested nutritional interventions that can improve muscle function and quality of life of the target group.

Purpose: The overall purpose is to investigate how muscle function and care-related quality of life can be maintained or improved through nutrition and physical activity interventions in older adults in nursing homes.

Study design and methods:

This cluster randomized controlled intervention study will be performed at six nursing homes in "Odsherred" City, Denmark. Participants and care staff from nursing homes will contribute to the design of this study protocol.

Sample size calculation:

Initially, the power calculation is performed by individual randomization based on the 30-second chair stand test. The starting point is six nursing homes are involved in the study. Approximately 40-50 residents are living in each location and assumable half of them want to participate in the project (n=20). A desired detectable change of 1.3, a P-value <0.05, and a power of 80%. The study has two arms (Usual care group (control) and nutritional and physical interventions group (intervention)) and the standardized difference in the nursing homes incl. intra cluster correlation, SD diff, nursing center = 0.42.

SD (diff., nursing center) =(SD (diff.,person))/√n, SD diff, person ≈1.87 If SD is 1.87 or less, the power will be at least 80% or greater. If there are more than 20 people per nursing home power will increase and if there are fewer than 20 people power will decrease.

Approximately 100 participants will be included and cluster randomized to either 12 months of collaborating developing (6 months) and testing (additional 6 months) nutritional and physical activity intervention (intervention group) or 12 months of usual care (control group). A simple random sample without replacement will be selected using the lottery method by statistical software (R).

Effects from the intervention will be examined by mixed methods that include both quantitative and qualitative data, as well as action research that focuses on creating development and change in collaboration with participants and care staff at the nursing homes.

Recruitment of participants and informed consent:

Recruitment of project participants takes place from "Odsherred" city's six nursing homes. The first step in recruitment takes place by the principal investigator orally and in writing informing the nursing homes, care staff, relatives, nursing home councils, and the residents of the nursing homes about the project's purpose, content, and course. In the next step, (oral information) the principal investigator, the care staff, and relatives talk to the residents. Participant information (written information) is provided. The written information contains a description of the project, its purpose, method, and possible consequences associated with the participant's participation.

In the trial, no serious adverse events or minor risks are expected. No biological materials are collected. A nurse at each of the nursing homes is included in the project and will be present during all data collection periods. The nurses will be involved immediately if any health issues or concerns about health issues should arise. This project meets the guidelines of the Declaration of Helsinki II, as well as the guidelines of the Regional Ethics Committee (EMN-2021-07672 ) and the University of Copenhagen Ethical Committee (504-0316/22-5000).

Participants have the opportunity to withdraw consent at any time during the project. If there are measurements, eg performance tests, which the participants do not want to participate in, available data is collected from the journaling system without participation in all measurements.

Data on participants who withdraw will be documented. Participants receive no fee or other benefits. Collection, storage, and processing of empirical data are done with the Danish Data Protection Agency's instructions for handling confidential information in research work of an empirical nature.

Nutritional and physical intervention:

The intervention is developed with a focus on nutritional needs and physical activities.

The Plan-Do-Study-Act (PDSA) model is used to redefine issues and relevant actions together with residents, care staff, nursing home management, and relatives. The intervention will be developed based on new knowledge from a descriptive pre-study, previous studies, practical experiences, the participant's experiences and wishes as well as the staff's experiences and wishes. In collaboration they will form an implementation catalog, from here, the nursing homes can select a relevant number of components, which will be tested and implemented in practice.

The development and implementation duration is 6 months and the PDSA model is repeated three times at two-month intervals to strengthen and qualify the intervention. The PDSA model is known to the city's staff in advance and is additionally used in connection to continuing education. In addition, everyday physical activities that contribute to maintaining/improving physical function are included, based on the potentials that are uncovered in the descriptive pre-study.

The development and implementation period was followed by testing the effects of the intervention components and 12 months follow-up data collection was performed.

Data collection:

Data are collected at baseline, after 6, and 12 months.

The primary outcome is sustained or improved muscle function, but other outcomes including the "Adult Social Care Outcomes Toolkit" (ASCOT) questionnaire, calf circumference, and nutritional risk using the Eating Validation Scheme (EVS) were also collected.

The data analysis takes into account that not all participants are included in all measurements.

Statistical analysis:

The analysis includes all data after randomization, regardless of non-compliance or lack of results.

The effect of measures and intervention is assessed using an analysis of covariates adjusted for potential confounders (sex and age), which will be used to compare the variables between groups.

The Fisher Xact Test or chi-square test will be used to compare groups of older adults with overnutrition in terms of body composition, muscle function, non-communicable disease, and nutritional risk.

Data on recruitment and participants' feasibility and compliance in relation to intervention will be assessed by descriptive and comparative analysis.

A statistical software program for scientific research "R" will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Living at the nursing homes in Odsherred City
* Informed consent form signed after receiving oral and written information
* Read, speak and understand Danish

Exclusion Criteria:

* Terminal ill

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength (HGS) | Baseline
  Muscle function assessed by HGS in kilograms as a unit. To measure HGS, the Standard Operating Procedure (SOP) was followed using a "Jamar Smart Hand Dynamometer". Three measurements on each hand will be completed, when participants were sitting upright and with the arm at a 90-degree angle.
  The test was performed by the principal researcher and trained clinical dietician students.
Change in Hand Grip Strength (HGS) | 6 months follow-up
  Muscle function assessed by HGS in kilograms as a unit. To measure HGS, the Standard Operating Procedure (SOP) was followed using a ¨"Jamar Smart Hand Dynamometer". Three measurements on each hand will be completed, when participants were sitting upright and with the arm at a 90-degree angle.
  The test was performed by the principal researcher and trained clinical dietician students.
Change in Hand Grip Strength (HGS) | 12 months follow-up
  Muscle function assessed by HGS in kilograms as a unit. To measure HGS, the Standard Operating Procedure (SOP) was followed using a ¨"Jamar Smart Hand Dynamometer". Three measurements on each hand will be completed, when participants were sitting upright and with the arm at a 90-degree angle.
  The test was performed by the principal researcher and trained clinical dietician students.
Chair Stand Test (CST) - 30 Second | Baseline
  Muscle function assessed by CST. The test requires the participant to stand up and sit down as many times as possible within 30 seconds according to Standard Operating Procedure (SOP). The participants are seated in a standard chair with their feet shoulder length apart and one foot in front of the other, doing as many stands as possible within 30 seconds. The unit is the number of full stands performed.
  Trained clinical dietician students and primary researcher will perform all tests
Change in Chair Stand Test (CST) - 30 Second | 6 months follow-up
  Muscle function assessed by CST. The test requires the participant to stand up and sit down as many times as possible within 30 seconds according to Standard Operating Procedure (SOP). The participants are seated in a standard chair with their feet shoulder length apart and one foot in front of the other, doing as many stands as possible within 30 seconds. The unit is the number of full stands performed.
  Trained clinical dietician students and primary researcher will perform all tests
Change in Chair Stand Test (CST) - 30 Second | 12 months follow-up
  Muscle function assessed by CST. The test requires the participant to stand up and sit down as many times as possible within 30 seconds according to Standard Operating Procedure (SOP). The participants are seated in a standard chair with their feet shoulder length apart and one foot in front of the other, doing as many stands as possible within 30 seconds. The unit is the number of full stands performed.
  Trained clinical dietician students and primary researcher will perform all tests

SECONDARY OUTCOMES:
Quality of Life by Adult Social Care Outcomes Toolkit (ASCOT) | Baseline
  Quality of life will be assessed by the Adult Social Care Outcomes Toolkit (ASCOT) questionnaire performed as an interview. The interview was performed by the principal researcher and trained clinical dietician students. The questionnaire ask the participants to give their own subjective evaluation of their experience for each of the eight domains including; Control over daily life, Personal cleanliness and comfort, Meals and nutrition, Safety, Social participation, Activities/occupation, Home cleanliness and comfort, and Dignity and respect.
  These subjective measures relate directly to the participant's capabilities i.e. the extent to which their experienced physical and physiological environment allows the participants to choose their own situations. The satisfaction was scaled from 'Very satisfied', 'Quite satisfied', 'Neither satisfied nor dissatisfied', to 'Quite or very dissatisfied' and 'Don't know'
Change in Quality of Life by Adult Social Care Outcomes Toolkit (ASCOT) | 6 months follow-up
  Quality of life will be assessed by the Adult Social Care Outcomes Toolkit (ASCOT) questionnaire performed as an interview. The interview was performed by the principal researcher and trained clinical dietician students. The questionnaire ask the participants to give their own subjective evaluation of their experience for each of the eight domains including; Control over daily life, Personal cleanliness and comfort, Meals and nutrition, Safety, Social participation, Activities/occupation, Home cleanliness and comfort, and Dignity and respect.
  These subjective measures relate directly to the participant's capabilities i.e. the extent to which their experienced physical and physiological environment allows the participants to choose their own situations.The satisfaction was scaled from 'Very satisfied', 'Quite satisfied', 'Neither satisfied nor dissatisfied', to 'Quite or very dissatisfied' and 'Don't know'
Change in Quality of Life by Adult Social Care Outcomes Toolkit (ASCOT) | 12 months follow-up
  Quality of life will be assessed by the Adult Social Care Outcomes Toolkit (ASCOT) questionnaire performed as an interview. The interview was performed by the principal researcher and trained clinical dietician students. The questionnaire ask the participants to give their own subjective evaluation of their experience for each of the eight domains including; Control over daily life, Personal cleanliness and comfort, Meals and nutrition, Safety, Social participation, Activities/occupation, Home cleanliness and comfort, and Dignity and respect.
  These subjective measures relate directly to the participant's capabilities i.e. the extent to which their experienced physical and physiological environment allows the participants to choose their own situations.The satisfaction was scaled from 'Very satisfied', 'Quite satisfied', 'Neither satisfied nor dissatisfied', to 'Quite or very dissatisfied' and 'Don't know'
Weight in kilograms | Baseline
  Weight is measured on a calibrated chair scale in the morning before breakfast. Participants are not wearing shoes and are dressed in light clothing. The units are in kilograms (kg).
  Changes in weight are assessed together with changes in Body Mass Index calculated by kg divided by height (m)^2
Change in weight in kilograms | 6 months follow-up
  Weight is measured on a calibrated chair scale in the morning before breakfast. Participants are not wearing shoes and are dressed in light clothing. The units are in kilograms (kg).
  Changes in weight are assessed together with changes in Body Mass Index calculated by kg divided by height (m)^2
Change in weight in kilograms | 12 months follow-up
  Weight is measured on a calibrated chair scale in the morning before breakfast. Participants are not wearing shoes and are dressed in light clothing. The units are in kilograms (kg).
  Changes in weight are assessed together with changes in Body Mass Index calculated by kg divided by height (m)^2

OTHER OUTCOMES:
Height in meters | Baseline
  Height will be measured on a stadiometer on participants that are able to stand.
  The unit is in meters (m). The participants will be measured without shoes and standing as straight as possible against the stadiometer.
  For participants not able to stand, height will be estimated by measuring the ulna in centimeters.
  The participants must bend the left arm with the palm across the chest and the fingers pointing towards the opposite shoulder. The distance between the point of the elbow (olecranon process) and the center of the prominent bone of the wrist (styloid process) are measured with a non-elastic tape.
  Height is measured for the purpose of estimating Body Mass Index (BMI).
  The test was performed by the principal researcher and trained clinical dietician students.
Calf circumference | Baseline
  When measuring the calf muscle, a non-elastic but flexible measuring tape is used.
  It must be able to measure around the calf muscle. The calf muscle is measured at the thickest point / largest circumference according to Standard Operating Procedure (SOP). The units are in centimeters.
  The test was performed by the principal researcher and trained clinical dietician students.
Change in calf circumference | 6 months follow-up
  When measuring the calf muscle, a non-elastic but flexible measuring tape is used.
  It must be able to measure around the calf muscle. The units are in centimeters.
  The test was performed by the principal researcher and trained clinical dietician students.
  The calf muscle is measured at the thickest point / largest circumference according to Standard Operating Procedure (SOP).
Change in calf circumference | 12 months follow-up
  When measuring the calf muscle, a non-elastic but flexible measuring tape is used.
  It must be able to measure around the calf muscle. The units are in centimeters.
  The test was performed by the principal researcher and trained clinical dietician students.
  The calf muscle is measured at the thickest point / largest circumference according to Standard Operating Procedure (SOP).
Nutritional risk | Baseline
  First participants will be assessed by the Eating Validation Scheme (EVS).The EVS assesses nutritional risk into three scores; 1) 'No risk', 2) 'risk of malnutrition', and 3) 'benefit from a nutritional intervention'.
  The test was performed by the principal researcher and trained clinical dietician students.
Change in nutritional risk | 6 months follow-up
  First participants will be assessed by the Eating Validation Scheme (EVS). The EVS assesses nutritional risk into three scores; 1) 'No risk', 2) 'risk of malnutrition', and 3) 'benefit from a nutritional intervention'.
  The test was performed by the principal researcher and trained clinical dietician students.
Change in nutritional risk | 12 months follow-up
  First participants will be assessed by the Eating Validation Scheme (EVS). The EVS assesses nutritional risk into three scores; 1) 'No risk', 2) 'risk of malnutrition', and 3) 'benefit from a nutritional intervention'.
  The test was performed by the principal researcher and trained clinical dietician students.

CONTACTS AND LOCATIONS:
Overall Officials: Margit AD Aaslyng, Ph.D., Study Chair — University College Absalon; Inge Tetens, Professor, Study Chair — University of Copenhagen; Anne Marie Beck, Master, Study Chair — Herlev and Gentofte University Hospital,Denmark; Anja W Dynesen, Ph.D., Study Chair — University College Absalon
Locations (6):
- Denmark (6):
  - Bobjerg Nursing Home, Asnæs, Region Sjælland
  - Grevinge Nusing Home, Grevinge, Region Sjælland
  - Solvognen Nursing home, Højby, Region Sjælland
  - Bakkegården Nursing home, Hørve, Region Sjælland
  - Grønnegården Nursing home, Nykøbing Sjælland, Region Sjælland
  - Præstevænget Nursing Home, Nykøbing Sjælland, Region Sjælland

IPD SHARING:
Plan to Share IPD: No
After study is finished, no data will be shared

REFERENCES:
- [Background] Beard JR, Officer A, de Carvalho IA, Sadana R, Pot AM, Michel JP, Lloyd-Sherlock P, Epping-Jordan JE, Peeters GMEEG, Mahanani WR, Thiyagarajan JA, Chatterji S. The World report on ageing and health: a policy framework for healthy ageing. Lancet. 2016 May 21;387(10033):2145-2154. doi: 10.1016/S0140-6736(15)00516-4. Epub 2015 Oct 29. PMID 26520231
- [Background] DiMilia PR, Mittman AC, Batsis JA. Benefit-to-Risk Balance of Weight Loss Interventions in Older Adults with Obesity. Curr Diab Rep. 2019 Nov 4;19(11):114. doi: 10.1007/s11892-019-1249-8. PMID 31686230
- [Background] Haywood CJ, Prendergast LA, Purcell K, Le Fevre L, Lim WK, Galea M, Proietto J. Very Low Calorie Diets for Weight Loss in Obese Older Adults-A Randomized Trial. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):59-65. doi: 10.1093/gerona/glx012. PMID 28329121
- [Background] Bouchonville MF, Villareal DT. Sarcopenic obesity: how do we treat it? Curr Opin Endocrinol Diabetes Obes. 2013 Oct;20(5):412-9. doi: 10.1097/01.med.0000433071.11466.7f. PMID 23974769
- [Background] Locher JL, Goldsby TU, Goss AM, Kilgore ML, Gower B, Ard JD. Calorie restriction in overweight older adults: Do benefits exceed potential risks? Exp Gerontol. 2016 Dec 15;86:4-13. doi: 10.1016/j.exger.2016.03.009. Epub 2016 Mar 17. PMID 26994938
- [Background] Goisser S, Kemmler W, Porzel S, Volkert D, Sieber CC, Bollheimer LC, Freiberger E. Sarcopenic obesity and complex interventions with nutrition and exercise in community-dwelling older persons--a narrative review. Clin Interv Aging. 2015 Aug 6;10:1267-82. doi: 10.2147/CIA.S82454. eCollection 2015. PMID 26346071
- [Background] Ard JD, Cook M, Rushing J, Frain A, Beavers K, Miller G, Miller ME, Nicklas B. Impact on weight and physical function of intensive medical weight loss in older adults with stage II and III obesity. Obesity (Silver Spring). 2016 Sep;24(9):1861-6. doi: 10.1002/oby.21569. Epub 2016 Jul 19. PMID 27430587
- [Background] Ard JD, Gower B, Hunter G, Ritchie CS, Roth DL, Goss A, Wingo BC, Bodner EV, Brown CJ, Bryan D, Buys DR, Haas MC, Keita AD, Flagg LA, Williams CP, Locher JL. Effects of Calorie Restriction in Obese Older Adults: The CROSSROADS Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2017 Dec 12;73(1):73-80. doi: 10.1093/gerona/glw237. PMID 28003374
- [Background] Beavers KM, Nesbit BA, Kiel JR, Sheedy JL, Arterburn LM, Collins AE, Ford SA, Henderson RM, Coleman CD, Beavers DP. Effect of an Energy-Restricted, Nutritionally Complete, Higher Protein Meal Plan on Body Composition and Mobility in Older Adults With Obesity: A Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2019 May 16;74(6):929-935. doi: 10.1093/gerona/gly146. PMID 30629126
- [Background] Frimel TN, Sinacore DR, Villareal DT. Exercise attenuates the weight-loss-induced reduction in muscle mass in frail obese older adults. Med Sci Sports Exerc. 2008 Jul;40(7):1213-9. doi: 10.1249/MSS.0b013e31816a85ce. PMID 18580399
- [Background] Kelly KR, Haus JM, Solomon TP, Patrick-Melin AJ, Cook M, Rocco M, Barkoukis H, Kirwan JP. A low-glycemic index diet and exercise intervention reduces TNF(alpha) in isolated mononuclear cells of older, obese adults. J Nutr. 2011 Jun;141(6):1089-94. doi: 10.3945/jn.111.139964. Epub 2011 Apr 27. PMID 21525252
- [Background] Muscariello E, Nasti G, Siervo M, Di Maro M, Lapi D, D'Addio G, Colantuoni A. Dietary protein intake in sarcopenic obese older women. Clin Interv Aging. 2016 Feb 5;11:133-40. doi: 10.2147/CIA.S96017. eCollection 2016. PMID 26917955
- [Background] Nicklas BJ, Brinkley TE, Houston DK, Lyles MF, Hugenschmidt CE, Beavers KM, Leng X. Effects of Caloric Restriction on Cardiorespiratory Fitness, Fatigue, and Disability Responses to Aerobic Exercise in Older Adults With Obesity: A Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2019 Jun 18;74(7):1084-1090. doi: 10.1093/gerona/gly159. PMID 29982294
- [Background] Waters DL, Vawter R, Qualls C, Chode S, Armamento-Villareal R, Villareal DT. Long-term maintenance of weight loss after lifestyle intervention in frail, obese older adults. J Nutr Health Aging. 2013 Jan;17(1):3-7. doi: 10.1007/s12603-012-0421-5. PMID 23299370
- [Background] Villareal DT, Shah K, Banks MR, Sinacore DR, Klein S. Effect of weight loss and exercise therapy on bone metabolism and mass in obese older adults: a one-year randomized controlled trial. J Clin Endocrinol Metab. 2008 Jun;93(6):2181-7. doi: 10.1210/jc.2007-1473. Epub 2008 Mar 25. PMID 18364384
- [Background] Villareal DT, Banks M, Sinacore DR, Siener C, Klein S. Effect of weight loss and exercise on frailty in obese older adults. Arch Intern Med. 2006 Apr 24;166(8):860-6. doi: 10.1001/archinte.166.8.860. PMID 16636211
- [Background] Villareal DT, Aguirre L, Gurney AB, Waters DL, Sinacore DR, Colombo E, Armamento-Villareal R, Qualls C. Aerobic or Resistance Exercise, or Both, in Dieting Obese Older Adults. N Engl J Med. 2017 May 18;376(20):1943-1955. doi: 10.1056/NEJMoa1616338. PMID 28514618
- [Background] Villareal DT, Miller BV 3rd, Banks M, Fontana L, Sinacore DR, Klein S. Effect of lifestyle intervention on metabolic coronary heart disease risk factors in obese older adults. Am J Clin Nutr. 2006 Dec;84(6):1317-23. doi: 10.1093/ajcn/84.6.1317. PMID 17158411
- [Background] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Netten A, Burge P, Malley J, Potoglou D, Towers AM, Brazier J, Flynn T, Forder J, Wall B. Outcomes of social care for adults: developing a preference-weighted measure. Health Technol Assess. 2012;16(16):1-166. doi: 10.3310/hta16160. PMID 22459668
- [Background] Landi F, Onder G, Russo A, Liperoti R, Tosato M, Martone AM, Capoluongo E, Bernabei R. Calf circumference, frailty and physical performance among older adults living in the community. Clin Nutr. 2014 Jun;33(3):539-44. doi: 10.1016/j.clnu.2013.07.013. Epub 2013 Jul 31. PMID 23948128
- [Background] Beck AM, Beermann T, Kjaer S, Rasmussen HH. Ability of different screening tools to predict positive effect on nutritional intervention among the elderly in primary health care. Nutrition. 2013 Jul-Aug;29(7-8):993-9. doi: 10.1016/j.nut.2013.01.016. Epub 2013 May 2. PMID 23644011
- [Background] Cederholm T, Bosaeus I, Barazzoni R, Bauer J, Van Gossum A, Klek S, Muscaritoli M, Nyulasi I, Ockenga J, Schneider SM, de van der Schueren MA, Singer P. Diagnostic criteria for malnutrition - An ESPEN Consensus Statement. Clin Nutr. 2015 Jun;34(3):335-40. doi: 10.1016/j.clnu.2015.03.001. Epub 2015 Mar 9. PMID 25799486
- [Background] Barbosa VM, Stratton RJ, Lafuente E, Elia M. Ulna length to predict height in English and Portuguese patient populations. Eur J Clin Nutr. 2012 Feb;66(2):209-15. doi: 10.1038/ejcn.2011.177. Epub 2011 Oct 12. PMID 21989325
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Barazzoni R, Jensen GL, Correia MITD, Gonzalez MC, Higashiguchi T, Shi HP, Bischoff SC, Boirie Y, Carrasco F, Cruz-Jentoft A, Fuchs-Tarlovsky V, Fukushima R, Heymsfield S, Mourtzakis M, Muscaritoli M, Norman K, Nyulasi I, Pisprasert V, Prado C, de van der Schuren M, Yoshida S, Yu Y, Cederholm T, Compher C. Guidance for assessment of the muscle mass phenotypic criterion for the Global Leadership Initiative on Malnutrition (GLIM) diagnosis of malnutrition. Clin Nutr. 2022 Jun;41(6):1425-1433. doi: 10.1016/j.clnu.2022.02.001. Epub 2022 Apr 19. PMID 35450768
- See also: Reference 2 — https://www.kl.dk/nyheder/makro-analyseenheden/nyt-om-dansk-oekonomi/ny-befolkningsfremskrivning-2020-2060/
- See also: Reference 3 — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight
- See also: Reference 32 — https://vbn.aau.dk/en/publications/omsorgsbetinget-livskvalitet-og-hjemmehjælp-en-ascot-undersøgelse
- See also: Reference 33 — https://apps.who.int/iris/bitstream/handle/10665/43392/924159392X_eng.pdf
- See also: Reference 34 — https://www.datatilsynet.dk/media/7753/danish-data-protection-act.pdf

DOCUMENTS (1):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT05804019/Prot_000.pdf